CLINICAL TRIAL: NCT00946452
Title: Symbicort SMART Satisfaction From Patient Perspective 2009
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-RMY-SYM-2009/1
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Asthma
Keywords: Control; Satisfaction
MeSH Terms: conditions — Asthma; Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To characterize the level of asthma control and patient satisfaction amongst diagnosed asthma sufferers who are currently receiving Symbicort Maintenance and Reliever Therapy (SMART) in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Have been prescribed Symbicort SMART (1 or 2 inhalation twice daily) by their Dr's for the past 3 months
* Informed consent

Exclusion Criteria:

* Symbicort SMART treatment < 3 months
* Patients requiring short courses of oral steroids more than twice in a month

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Score level of Satisfaction in Asthma Treatment Questionnaire (SATQ) | After 3 months on SMART - once
Score level of Asthma Control Test (ACT) | After 3 months on SMART - once

CONTACTS AND LOCATIONS:
Overall Officials: Liam Chong Kin, Professor, Principal Investigator — UMMC
Locations (1):
- Research Site, Petaling Jaya, Selangor, Malaysia